CLINICAL TRIAL: NCT02569008
Title: Study of Changes on Mean Systemic Filling Pressure (Pmsf) in Post-surgical Patients After a Fluid Challenge: Looking for the Minimal Dose of Fluids
Brief Title: Minimal Volume for Fluid Challenge in Post-operative Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 13.0116
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Post Cardiac Surgery
Keywords: Fluid Challenge; Mean systemic filling pressure; Fluid therapy
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 ml / Kg (Experimental): Patients receive a Fluid challenge with Compound Sodium Lactate 1 ml/Kg IV over 5 minutes
  Interventions: Drug: Fluid challenge with Compound Sodium Lactate
- 2 ml/Kg (Experimental): Patients receive a Fluid challenge with Compound Sodium Lactate 2 ml/Kg IV over 5 minutes
  Interventions: Drug: Fluid challenge with Compound Sodium Lactate
- 3 ml/Kg (Experimental): Patients receive a Fluid challenge with Compound Sodium Lactate 3 ml/Kg IV over 5 minutes
  Interventions: Drug: Fluid challenge with Compound Sodium Lactate
- 4 ml/Kg (Experimental): Patients receive a Fluid challenge with Compound Sodium Lactate 4 ml/Kg IV over 5 minutes
  Interventions: Drug: Fluid challenge with Compound Sodium Lactate

INTERVENTIONS:
Drug: Fluid challenge with Compound Sodium Lactate — Infusion of the mentioned dose of Compound sodium Lactate over 5 minutes intravenously.
  Other Names: Hartmann's Solution

SUMMARY:
This study evaluate the effect of different doses of crystalloids on the changes on cardiac output (CO) and on the proportion of responders and non-responders and aims to determine the minimal volume required to increase the mean systemic filling pressures (Pmsf) in post-cardiac surgical patients.

DETAILED DESCRIPTION:
OBJECTIVES

1. To determine if different doses of fluids in a fluid challenge affect the change in CO and the proportion of responders / non-responders
2. To determine the minimal amount of volume required for performing an effective fluid challenge.

   1. To define the least significant change of the Pmsf measured by Pmsf-arm.
   2. To define the stop-flow time required to measure Pmsf-arm
3. To study the changes generated by a fluid challenge in the microcirculation and correlate those changes with the changes in the Pmsf.

STUDY DESIGN

1. TYPE OF STUDY This is an quasi-randomised open-label study. The purpose of this study is non-commercial.
2. STUDY OF MINIMAL VOLUME Once the participant is admitted to the ICU, and the monitors are in place, the fluid challenge will be administered. Each fluid challenge will be administered with a syringe (50 ml) in five minutes. In order to observe the effect of the volume on Pmsf-arm, the total sample of patients will be divided in 4 groups: in group one Pmsf-arm will be measured at baseline and after 1 ml/kg of body weight; in group 2 after 2 ml/Kg; in group 3 after 3 ml/kg and finally in group 4 after 4 ml/Kg. The fluid challenge will be completed in everybody after the measurement of Pmsf-arm, in order to respect clinical practice. Pmsa will be observed also. The total duration of the fluid challenge will be 5 minutes. The fluid challenge will be repeated in accordance with the clinical protocol or with the clinician advice.

   The first 20 patients will receive 4 ml/kg (normal clinical practice) between the base line and the second measurement of Pmsf-arm. The subsequent 20 patients will receive 3ml/kg between the two measurements of Pmsf-arm, and then 1ml/kg will be added to complete the normal fluid challenge. The following 20 patients will receive 2 ml/Kg between the two measurement of Pmsf-arm, and then the remaining 2 ml/kg will be given to complete the normal fluid challenge. And finally, the last 20 patients will receive 1 ml/kg between the two measurements of Pmsf-arm, and 3 ml/kg will be added to complete clinical practice.
3. STUDY OF MICROCIRCULATION In 25 patients, functional capillary density (FCD) microvascular flow index (MFI), proportion of perfused vessels (PPV) and microvascular heterogeneity index (MHI) will be measured with a side-stream dark-field (SDF) camera at five time points: (1)Baseline, (2) At the end of the fluid challenge (4 ml / kg in 5 minutes), (3) 5 minutes after the end of the fluid challenge, (4) 10 minutes after the end of the fluid challenge, (5) 15 minutes after the end of the fluid challenge.

   The ventilation settings, sedation and vasoactive support will be kept constant during the study period, unless other clinical instruction, in which case the data will be excluded from the analysis.
4. HAEMODYNAMIC MEASUREMENTS

4.1 CLINICAL MONITORING These measurements are using normally in clinical practice and will be used during the study but do not constitute any change in clinical practice.

* Mean arterial pressure (MAP) will be measured with a radial artery catheter (p.e. 115.090 Vygon, Ecouen, France).
* Central venous pressure (CVP) will be measured with a venous central catheter (p.e. CV-15854, Arrow International, Reading, USA) inserted in the internal jugular vein or the subclavian vein. This line will be ideally inserted in the anaesthetic room after induction of general anaesthesia. Once the study finishes, this line will be removed unless the clinical team taking care of the patient decided to use it.
* Both catheters will be connected to a pressure transducer (T001650A, Edwards Lifesciences LLC, Irvine, USA) and to a multi-parameter monitor (InfinityTM Delta, Dragger Medical Systems, USA). Zero levels of blood pressures were referenced to the intersection of the anterior axillary line and the fifth intercostal space.
* Cardiac output will be monitored using LiDCO TM plus (LiDCO Ltd, Cambridge, UK)

4.2 DETERMINATION OF PMSF-ARM Pmsf can be estimated measuring the venous pressure (Pv) and the arterial pressure (Pa) in on limb after rapid vascular occlusion. This estimation assumes Pa and Pv equilibrium following a rapid vascular occlusion as described by Maas et al[2]. In order to determine stop-flow time (or time of arterial / venous balance), we will perform a pilot study in 10 patients. We will measure the radial arterial pressure and venous pressure in the same hand and we will then stop the blood-ﬂow during 30 -60 seconds using an automatic pneumatic tourniquet (APT pneumatic tourniquet, Anetic Aid, Ltd. Guiseley, UK) to pressures 50 mmHg above systolic pressure. Measures will be taken three times in order to assess repeatability. The time required to equilibrate arterial and venous pressure will be the stop-flow time, and will be the time that we need to wait with the tourniquet inflated. In Maas study was between 25 - 30 seconds.

4.3 MICROCIRCULATION MEASUREMENTS

In order to study microcirculatory changes, sublingual microcirculatory videos will be obtained using a side-stream dark field-imaging device (SDF; Microscan, MicroVissionMedical, Amsterdam, the Nederlands) derived from the orthogonal polarized spectral imaging technology. Images acquisition and analysis will be performed according international recommendations [3] with dedicated software analysis (Automated Vascular Analysis (AVA) v. 1.0; Academic Medical Center, University of Amsterdam, Amsterdam, the Nederlands). These recommendations are summarised below:

* Image acquisition will include five sublingual good quality sequences of 20 seconds each at every observation time-point.
* Scoring will include measurement of perfused capillary density and evaluation of heterogeneity. We will measure:

  1. Functional capillary density (FCD): this can be calculated counting the number of intersection of capillaries with arbitrary grid lines and measurement of total capillary length relative to image area.
  2. Microcirculatory flow index (MFI): this is based on determination of the predominant type of flow in four quadrants. Flow is characterised as absent (0), intermittent (1), sluggish (2) or normal (3). The values of the four quadrants is averaged.
  3. Proportion of perfused vessels (PPV %): calculated as the total number of vessels minus the number of vessels with intermittent flow or no flow divided by the total number of vessels.
  4. Flow heterogeneity index (FHI): the difference between the highest MFI minus the lowest site MFI divided by the mean flow velocity of all sublingual sites at a single time point.

SETTING General and cardiothoracic intensive care unit, St George's Healthcare Trust.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the general or cardiothoracic intensive care unit, requiring fluid therapy guided by the current clinical protocol.

Exclusion Criteria:

* Extensive peripheral arterial occlusive disease in upper limbs.
* Postoperative valvular insufficiency
* Aortic valve regurgitation
* Arrhythmia
* Cardiac assist device (Intra-Aortic balloon pump)
* Right ventricular failure
* Patients without capacity to consent for themselves Also, patients requiring aggressive fluid resuscitation due to life-threatening cardiovascular instability and pregnant women will be excluded from the study.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Proportion of Responders by dose group | 15 minutes
  Proportion of responders to a fluid challenge by dose of crystalloids according to CO response (greater than 10% change in CO is a positive response)

SECONDARY OUTCOMES:
Change in Pmsf by dose of fluids | 15 Minutes
  change in Pmsf achieved by each group adjusted by baseline values
Minimal dose of fluids | 15 Minutes
  Estimated minimal dose of fluids required to achieve a significant change in Pmsf

CONTACTS AND LOCATIONS:
Overall Officials: Hollmann D Aya, M.D., Principal Investigator — St George's University Hospitals NHS Foundation Trust; Maurizio Cecconi, MD(Res), Study Director — St George's University Hospitals NHS Foundation Trust
Locations (1):
- St George's University Hospitals, NHS Foundation Trust, London, London, United Kingdom